CLINICAL TRIAL: NCT04386512
Title: Épidémiologie Clinique et caractéristiques Des Cas de Covid-19 Survenus Dans un Contexte de Lymphome Lors de la première Phase épidémique
Brief Title: Clinical Epidemiology and Characteristics Of Covid-19 Cases Occurred In A Lymphoma Setting In The First Epidemic Phase (LymphoCov1)
Acronym: LymphoCov1
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Caroline BESSON, investigator MD, Versailles Hospital
Other Study IDs: P20/12_LymphoCov
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: COVID; Lymphoma
Keywords: covid; lymphoma; epidemiology
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this retrospective clinical epidemiology study is to describe the characteristics of Covid-19 cases requiring hospitalization in adult patients with lymphomas during the initial phase of the epidemic (from 01/03/20 to 30/04/20).

The specific objectives are to estimate the frequency of severe forms of Covid-19 and those requiring intensive care hospitalisation, as well as the mortality related to the epidemic among the active file of patients followed for lymphoma at each study site, to investigate whether certain chemotherapy and/or immunotherapy treatments seem to be associated with severe forms or prolonged evolutions of Covid-19, to describe possible atypical clinical forms among the population of patients treated for lymphoma.

Translated with www.DeepL.com/Translator (free version)

DETAILED DESCRIPTION:
I

Methods :

* Multicentric retrospective observational epidemiological study based on the collection of data from patient records.
* Selection of voluntary hospital sites in regions with excess mortality during the epidemic phase.
* Systematic identification of Covid-19 cases from coding data (PMSI) from the medical information departments which will be compared with the numbers of patients followed for lymphoma in the haematology departments of each site during the 6 months preceding the epidemic, identified through the PMSI.
* Establishment of an ad hoc CRF for cases only with collection of clinical data concerning lymphoma and Covid-19 and routine biological data: Cytopenia (and in particular depth of lymphopenia), hypogammaglobulinemia, inflammatory markers.
* Estimated total number of sites: 10-15 and number of cases to be collected: 50-60.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age with lymphoma and a diagnosis of Covid-19 requiring hospitalization.
* In order not to bias the data by excluding patients with adverse outcomes, we will also collect data from deceased patients.

Exclusion Criteria:

Patients who refused to participate

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a current or past history of lymphoma who were hospitalized with Covid-19 infection between March the 1st and April the 30th in ile de France or Est region in France
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
mortality | 2 months
transfer to ICU | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Versailles, Le Chesnay, France